CLINICAL TRIAL: NCT05889767
Title: Indicators of Gut Permeability in Normal-weight Obesity in Response to Brief, Maximal and Sustained, Submaximal Exercise
Brief Title: Exercise-Induced Gut Permeability in Normal-weight Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oklahoma State University (Other)
Responsible Party: Principal Investigator, Sam Emerson, Associate Professor of Nutritional Sciences, Oklahoma State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-22-28-STW
Record Dates: First submitted 2023-05-04; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Normal-weight Obesity; Obesity
MeSH Terms: conditions — Obesity | interventions — Exercise Test

STUDY DESIGN:
Intervention Model Description: Three study groups (n=10/ group):
  1. Normal weight and low body fat percent (BMI 18.5-24.9 kg/m2, body fat percent < 25% in males or < 35% in females),
  2. Normal-weight obesity (BMI 18.5-24.9 kg/m2, body fat percent > 25% in males or > 35% in female)
  3. Overt obesity and high body fat percent (BMI > 30 kg/m2, body fat percent > 25% in males or > 35% in females)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal weight and low body fat percent (Active Comparator): The low risk comparator group for this study will consist of individuals with normal BMI (18.5 - 24.9 kg/m2) and body fat percent < 25% (male) or < 35% (female).
  Interventions: Other: Exercise tests (VO2 max test and 45-minute exercise session at 65% VO2 max)
- Normal-weight obesity (Experimental): Individuals with normal-weight obesity will be defined as having normal BMI (18.5 - 24.9 kg/m2), body fat percent > 25% (male) or > 35% (female).
  Interventions: Other: Exercise tests (VO2 max test and 45-minute exercise session at 65% VO2 max)
- Overt obesity and high body fat percent (Active Comparator): Overt obesity (BMI > 30 kg/m2) with high body fat percent (> 25% [male] or > 35% [female]) will be used as a high-risk comparator group.
  Interventions: Other: Exercise tests (VO2 max test and 45-minute exercise session at 65% VO2 max)

INTERVENTIONS:
Other: Exercise tests (VO2 max test and 45-minute exercise session at 65% VO2 max) — All participants will complete two exercise sessions:
  1. VO2 max test on a cycle ergometer
  2. Moderate exercise session (45 minutes at 65% measured VO2 max)

SUMMARY:
Exercise acutely increases gut permeability and inflammation, even in healthy populations. However, whether this response differs in groups at-risk for CVD that present with low-grade inflammation (e.g., normal-weight obesity) has yet to be examined. The investigators aim to measure serum indicators of gut permeability in those with normal-weight obesity pre- and post-short, intense exercise and sustained, moderate exercise

DETAILED DESCRIPTION:
The investigator's overall goal is to examine how indicators of gut permeability change in response to exercise in individuals with normal-weight obesity (i.e., normal body mass index [BMI] and high body fat percent) relative to those with a normal BMI and low body fat percent and those with a BMI in the obesity range and high body fat percent.

The investigators will examine indicators of gut permeability (specified in primary outcomes) in response to a short, intense bout of exercise (i.e., VO2 max test on a cycle ergometer) and sustained, moderate bout of exercise (i.e., 45 minutes at 65% measured VO2 max on a cycle ergometer).

Additionally, the investigators will measure basic anthropometrics, blood lipids and glucose, and body composition with DXA.

ELIGIBILITY:
Inclusion Criteria:

Control group: normal BMI, body fat percentage < 25% (male) or < 35% (female)

Normal-weight obesity: normal BMI, body fat percentage > 25% (male) or > 35% (female)

Overt obesity: BMI in obesity range, body fat percentage > 25% (male) or > 35% (female)

Exclusion Criteria:

* Presence of pacemaker
* Pregnant
* Postmenopausal status
* History of chronically using of tobacco products, illicit drugs, anti-inflammatory drugs (e.g., NSAIDs), lipid lowering drugs
* Recent use of antibiotics (< 6 weeks) and NSAIDs (< 3 days)
* Established cardiometabolic disease (e.g., cardiovascular disease, type 2 diabetes) diseases inflammatory in nature (e.g., rheumatoid arthritis, inflammatory bowel disease), and/or diagnosed irritable bowel syndrome.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Serum concentrations of FABP2 following short, intense exercise | Approximately 8 months
  The investigators will examine peak and absolute change in this indicator of gut permeability after the VO2 max test on a cycle ergometer.
Serum concentrations of LBP following short, intense exercise | Approximately 8 months
  The investigators will examine peak and absolute change in this indicator of gut permeability after the VO2 max test on a cycle ergometer.
Serum concentrations of sCD14 following short, intense exercise | Approximately 8 months
  The investigators will examine peak and absolute change in this indicator of gut permeability after the VO2 max test on a cycle ergometer.
Serum concentrations of FABP2 following sustained, moderate exercise | Approximately 8 months
  The investigators will examine peak and absolute change in this indicator of gut permeability after 45-minutes of exercise at 65% VO2 max on a cycle ergometer.
Serum concentrations of IL-6 following sustained, moderate exercise | Approximately 8 months
  The investigators will examine peak and absolute change in this inflammatory marker after 45-minutes of exercise at 65% VO2 max on a cycle ergometer.

SECONDARY OUTCOMES:
VO2 Max | Approximately 8 months
  The investigators will compare VO2 max after the short, intense exercise session across study groups.
Respiratory exchange ratio (RER) during VO2 max test | Approximately 8 months
  The investigators will compare RER dynamics during the short, intense exercise session across study groups.
Maximum workload during exercise sessions | Approximately 8 months
  The investigators will compare workload dynamics in watts during the short, intense and moderate, sustained exercise session across study groups.
Heart rate dynamics during exercise sessions | Approximately 8 months
  The investigators will compare heart rate dynamics during the short, intense and moderate, sustained exercise session across study groups.

OTHER OUTCOMES:
Body fat percent assessment with dual-energy X-ray absorptiometry (DXA). | Approximately 8 months
  The investigators will perform DXA scans on all participants to assess body fat percent.
Absolute body fat assessment with dual-energy X-ray absorptiometry (DXA) | Approximately 8 months
  The investigators will perform DXA scans on all participants to assess absolute body fat in kilograms.
Lean mass percent assessment with dual-energy X-ray absorptiometry (DXA) | Approximately 8 months
  The investigators will perform DXA scans on all participants to assess lean mass percent.
Absolute lean mass assessment with dual-energy X-ray absorptiometry (DXA) | Approximately 8 months
  The investigators will perform DXA scans on all participants to assess absolute lean mass in kilograms.
Absolute visceral fat mass assessment with dual-energy X-ray absorptiometry (DXA) | Approximately 8 months
  The investigators will perform DXA scans on all participants to assess absolute visceral mass in grams.
Lipid panel with Abbott Piccolo Xpress Clinical Chemistry Analyzer | Approximately 8 months
  The investigators will perform a lipid panel on all participants.

CONTACTS AND LOCATIONS:
Locations (1):
- 208 Nancy Randolph Davis, Oklahoma State University, Stillwater, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided